CLINICAL TRIAL: NCT03416374
Title: An Open-label, Single-Arm, Multicenter Study to Evaluate the Efficacy and Safety of Ixazomib in Combination With Lenalidomide and Dexamethasone in Patients With Relapsed and/or Refractory Multiple Myeloma Initially Treated With an Injection of Proteasome Inhibitor-Based Therapy
Brief Title: A Study to Evaluate the Efficacy and Safety of Ixazomib in Combination With Lenalidomide and Dexamethasone in Patients With Relapsed and/or Refractory Multiple Myeloma Initially Treated With an Injection of Proteasome Inhibitor-Based Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C16043; U1111-1207-0061 (Other: WHO); JapicCTI-183839 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2018-01-23; First posted 2018-01-31 (Actual); Results first posted 2022-08-22 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-05

CONDITIONS: Relapsed and/or Refractory Multiple Myeloma
MeSH Terms: interventions — ixazomib; Bortezomib; carfilzomib; Lenalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Combination Therapy + Ixazomib Therapy (Experimental): Bortezomib + Lenalidomide + Dexamethasone, or Carfilzomib + Lenalidomide + Dexamethasone, standard recommended dose according to the package insert of each drug (Treatment Period I), followed by Ixazomib (4.0 mg) on Days 1, 8 and 15, plus Lenalidomide (25 mg) on Days 1 to 21, and Dexamethasone (40 mg) on Days 1, 8, 15 and 22, of a 28-day cycle (Treatment Period II)
  Interventions: Drug: Ixazomib; Drug: Bortezomib; Drug: Carfilzomib; Drug: Lenalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Ixazomib — Ixazomib capsules
Drug: Bortezomib — Bortezomib injections
Drug: Carfilzomib — Carfilzomib intravenous infusions
Drug: Lenalidomide — Lenalidomide capsules
Drug: Dexamethasone — Dexamethasone tablets

SUMMARY:
The purpose of this study is to investigate the efficacy and safety of long-term administration of the oral proteasome inhibitor ixazomib as part of ixazomib in combination with lenalidomide and dexamethasone (IRd) therapy in patients with relapsed and/or refractory multiple myeloma (RRMM) treated initially with an injectable proteasome inhibitor-based therapy.

DETAILED DESCRIPTION:
The drug being tested in this study is called Ixazomib. Ixazomib is being tested to treat people who have RRMM. This study will look at the effectiveness and safety of IRd in participants with RRMM previously receiving an injectable proteasome inhibitor-based therapy. This study consists of two treatment periods, Treatment Period I and Treatment Period II.

The study will enroll 47 patients. All participants will receive following treatment:

- Combination therapy with Bortezomib + Lenalidomide + Dexamethasone (VRd) or combination therapy with Carfilzomib + Lenalidomide + Dexamethasone (KRd), standard recommended dose according to the package insert of each drug, as Treatment Period I, followed by Combination therapy with Ixazomib 4.0 mg + Lenalidomide 25 mg + Dexamethasone 40 mg (IRd) as Treatment Period II

At start of this study, combination therapy of VRd or KRd will be decided by investigator as Treatment Period I after the baseline evaluations. After the start of Treatment Period I, a participant's eligibility for Treatment Period II is then determined 3 cycles. Participants who meet these eligibility criteria II subsequently continue into Treatment Period II and receive IRd.

This multi-center trial will be conducted in Japan. It is anticipated that the treatment phase of this study will last up to 39 months, including 18 months for enrollment. Participants will make multiple visits to the clinic in treatment period, and follow-up period including a follow-up assessment after last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

Eligibility for Treatment Period I

1. Men and women of age 20 years or older at the time of enrollment.
2. Participants with RRMM.
3. Participants who are planned to start combination therapy with bortezomib, lenalidomide, and dexamethasone (VRd) or carfilzomib, lenalidomide, and dexamethasone (KRd) as second, third or fourth line of treatment.
4. Participants with measurable disease defined by one or more of the following three measurements.

   * Serum M-protein: ≥0.5 gram (g)/ deciliter (dL) (≥ 5 g/ liter [L])
   * Urine M-protein: ≥ 200 milligram (mg)/24 hours
   * Serum free light chain assay: involved free light chain concentration ≥ 10 mg/dL (≥ 100 mg/L) provided that the serum free light chain ratio is abnormal
5. Participants with Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-2; however, participants with ECOG PS 3 are eligible if they only have symptoms associated with bone lesions.
6. Participants who are considered by the principal investigator or investigator not to be eligible for transplant; or, if considered eligible for transplant, participants who are planned not to undergo transplant for at least 12 months after the start of the study treatment.
7. Participants must be registered with, and comply with, the guidelines of the lenalidomide management program.
8. Participants who, before implementing procedures related to clinical research (excluding standard medical practices), understand that they can withdraw consent at any time without suffering from disadvantages to future treatments, and can provide written informed consent.

   Eligibility for Treatment Period II
9. Participants must have received an injectable proteasome inhibitor (bortezomib or carfilzomib) in each treatment cycle of Treatment Period I.

Exclusion Criteria:

Eligibility for Treatment Period I

1. Women who are nursing or pregnant.
2. Participants with another active malignancy, i.e. synchronous active malignancy or previous malignancy with a disease-free period of less than 5 years, except for participants with carcinoma in situ (intraepithelial carcinoma) or intramucosal carcinoma judged to be cured by topical treatment.
3. Participants with poorly controlled active thrombosis.
4. Participants who have participated in a clinical trial of ixazomib or have been treated with ixazomib.
5. Participants who were refractory to either treatment regimen based on lenalidomide and/or proteasome inhibitor(s).

   Note: Refractory MM is defined as PD on therapy or PD within 60 days after the last dose of a given therapy. Participants who have disease progressed 60 days after the last dose of a given therapy will be considered as relapsed in this study.
6. Participants with ongoing or active systemic infection, known hepatitis B virus infection, known hepatitis C virus infection, or known positivity to human immunodeficiency virus (HIV).
7. Participants who underwent major surgery within 14 days prior to enrollment to Treatment Period I. Surgery for bone lesions is not considered as major surgery.
8. Participants who received radiation therapy within 14 days prior to enrollment to Treatment Period I. If the radiation field is small, 7 days is considered as a sufficient interval between radiation therapy and chemotherapy.
9. Participants who experience Grade 1 peripheral neuropathy accompanied by pain, or Grade ≥2 peripheral neuropathy.
10. Evidence of current uncontrolled cardiovascular conditions, including uncontrolled hypertension, uncontrolled cardiac arrhythmia, symptomatic congestive heart failure, unstable angina, or myocardial infarction within the past 6 months before enrollment to Treatment Period I.
11. Infection requiring systemic antibiotic therapy or other serious infection within 14 days before enrollment into Treatment Period I.
12. Participants with central nervous system involvement.
13. Inability to swallow oral medications, inability or unwillingness to comply with the drug administration requirements, or gastrointestinal conditions that could interfere with the oral absorption or tolerance of treatment.
14. Psychiatric illness/social situation that would limit compliance with study requirements.
15. Comorbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the participant inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens.

    Eligibility for Treatment Period II
16. Participants who do not achieve at least a minimal response (MR) to VRd or KRd in Treatment Period I per the International Myeloma Working Group (IMWG) response criteria, 2014 revision.
17. Participants who experience Grade 1 peripheral neuropathy accompanied by pain, or Grade ≥2 peripheral neuropathy during Treatment Period I.
18. Participants with evidence of uncontrolled cardiovascular conditions, including uncontrolled hypertension, uncontrolled cardiac arrhythmia, symptomatic congestive heart failure, unstable angina, or myocardial infarction during Treatment Period I.
19. Participants using potent CYP3A4 inducing agents (rifampicin, rifapentine, rifabutin, carbamazepine, phenytoin, phenobarbital), or gingko biloba or St. John's wort.
20. Participants with hypersensitivity to any of the IRd study medications, their analogs, or excipients contained in IRd.
21. Comorbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the participant inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2018-02-18 (Actual); Primary Completion 2021-05-28 (Actual); Study Completion 2021-05-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (23):
- Japan (23):
  - Kameda Medical Center, Kamogawa, Chiba
  - The Jikei University Kashiwa Hospital, Kashiwa, Chiba
  - Ogaki Municipal Hospital, Ōgaki, Gifu
  - Gunma University Hospital, Maebashi, Gunma
  - Shibukawa Medical Center, Shibukawa, Gunma
  - Kobe city Medical Center General Hospital, Kobe, Hyōgo
  - Kanazawa University Hospital, Kanazawa, Ishikawa-ken
  - Iwate Medical University, Morioka, Iwate
  - Yokohama Municipal Citizen's Hospital, Yokohama, Kanagawa
  - Suwa Red Cross Hospital, Suwa, Nagano
  - Dokkyo Medical University, Koshigaya, Saitama
  - Juntendo University Hospital, Bunkyo-ku, Tokyo
  - Nippon Medical School Hospital, Bunkyo-ku, Tokyo
  - Nihon University Itabashi Hospital, Itabashi-ku, Tokyo
  - The Cancer Institute Hospital of JFCR, Koto-ku, Tokyo
  - The Jikei University Hospital, Minato-ku, Tokyo
  - Kyorin University Hospital, Mitaka, Tokyo
  - Japanese Red Cross Medical Center, Shibuya-ku, Tokyo
  - Tokyo Disaster Medical Center, Tachikawa, Tokyo
  - Hiroshima Red Cross Hospital & Atomic-bomb Survivors Hospital, Hiroshima
  - Kyoto Kuramaguchi Medical Center, Kyoto
  - Niigata Cancer Center Hospital, Niigata
  - Osaka Red Cross Hospital, Osaka

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Abe Y, Sasaki M, Takezako N, Ito S, Suzuki K, Handa H, Chou T, Yoshida T, Mori I, Shinozaki T, Suzuki K. Efficacy and Safety of Ixazomib Plus Lenalidomide and Dexamethasone Following Injectable PI-Based Therapy in Relapsed/Refractory Multiple Myeloma. Ann Hematol. 2023 Sep;102(9):2493-2504. doi: 10.1007/s00277-023-05212-7. Epub 2023 Jun 21. PMID 37341778
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5f6b60204db2bf003ab49579

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participant s took part in the survey at 33 investigative sites in Japan, from 18 February 2018 to 28 May 2021.
Pre-assignment Details: A total of 45 participants were enrolled and received the study treatment in this study.
Groups:
- [VRd]; Bortezomib + Lenalidomide + Dexamethasone Therapy: Bortezomib + Lenalidomide + Dexamethasone, standard recommended dose according to the package insert of each drug (Treatment Period I), followed by Ixazomib (4.0 mg) on Days 1, 8 and 15, plus Lenalidomide (25 mg) on Days 1 to 21, and Dexamethasone (40 mg) on Days 1, 8, 15 and 22, of a 28-day cycle (Treatment Period II)
- [KRd]; Carfilzomib + Lenalidomide + Dexamethasone Therapy: Carfilzomib + Lenalidomide + Dexamethasone, standard recommended dose according to the package insert of each drug (Treatment Period I), followed by Ixazomib (4.0 mg) on Days 1, 8 and 15, plus Lenalidomide (25 mg) on Days 1 to 21, and Dexamethasone (40 mg) on Days 1, 8, 15 and 22, of a 28-day cycle (Treatment Period II)
Period: Treatment Period I
Arm/Group | [VRd]; Bortezomib + Lenalidomide + Dexamethasone Therapy | [KRd]; Carfilzomib + Lenalidomide + Dexamethasone Therapy
Started | 6 | 39
Completed | 0 | 0
Not Completed | 6 | 39
Period: Between Treatment Period I and II
Arm/Group | [VRd]; Bortezomib + Lenalidomide + Dexamethasone Therapy | [KRd]; Carfilzomib + Lenalidomide + Dexamethasone Therapy
Started | 6 | 39
Completed | 6 | 30
Not Completed | 0 | 9
Not completed — Other | 0 | 9
Period: Treatment Period II
Arm/Group | [VRd]; Bortezomib + Lenalidomide + Dexamethasone Therapy | [KRd]; Carfilzomib + Lenalidomide + Dexamethasone Therapy
Started | 6 | 30
Completed | 2 | 12
Not Completed | 4 | 18
Not completed — Lack of Efficacy | 3 | 11
Not completed — Adverse Event | 1 | 4
Not completed — Death | 0 | 1
Not completed — Other | 0 | 2

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): all participants who were enrolled in Treatment Period I and who receive at least one dose of any therapy during the Treatment Period.
Groups:
- Total: Total of all reporting groups
Arm/Group | [VRd]; Bortezomib + Lenalidomide + Dexamethasone Therapy | [KRd]; Carfilzomib + Lenalidomide + Dexamethasone Therapy | Total
Number analyzed (Participants) | 6 | 39 | 45
Age, Continuous [Mean (Standard Deviation); unit: Years] | 71.8 (8.57) | 70.5 (9.40) | 70.7 (9.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 16 | 21
  Male | 1 | 23 | 24
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants] — All participants were enrolled in Japan.
  Participants
    Japan | 6 | 39 | 45
Height [Mean (Standard Deviation); unit: Centimeters (cm)] | 153.0 (9.70) | 158.5 (8.29) | 157.8 (8.58)
Weight [Mean (Standard Deviation); unit: Kilograms (kg)] — Population: The number analyzed is the number of participants with data available for analysis.
  Kilograms (kg)
    number analyzed (Participants) | 6 | 37 | 43
    (all) | 52.85 (7.204) | 57.87 (10.380) | 57.17 (10.081)
BMI [Mean (Standard Deviation); unit: Kilogram (kg)/meter (m)^2]] — Body Mass Index = weight (kg)/[height (m)^2] Population: The number analyzed is the number of participants with data available for analysis.
  Kilogram (kg)/meter (m)^2]
    number analyzed (Participants) | 6 | 37 | 43
    (all) | 22.60 (2.619) | 22.91 (2.512) | 22.86 (2.497)
Body Surface Area [Mean (Standard Deviation); unit: m^2] — Population: The number analyzed is the number of participants with data available for analysis.
  m^2
    number analyzed (Participants) | 6 | 37 | 43
    (all) | 1.487 (0.1395) | 1.583 (0.1760) | 1.569 (0.1732)
International Staging System (at Initial Diagnosis) [Count of Participants; unit: Participants] — International Staging System is a staging system for cancer progression. Stages are classified by Stage I to Stage III. Stage I: Serum beta2-microglobulin <3.5 mg/L and albumin ≥3.5 g/dL; Stage II: Neither Stage I or III, meaning that either: beta2-microglobulin level ≥3.5 and <5.5 mg/L (with any albumin level), OR albumin <3.5 g/dL with beta2-microglobulin <3.5 mg/L; Stage III: Serum beta2-microglobulin ≥5.5 mg/L. Normal serum beta2-microglobulin: <3.0 mg/L; normal albumin: 3.5-5.0 g/dL.
  Participants
    Stage I | 2 | 17 | 19
    Stage II | 3 | 14 | 17
    Stage III | 1 | 8 | 9
International Staging System (at First Treatment [Period I]) [Count of Participants; unit: Participants]
  Stage I | 5 | 19 | 24
  Stage II | 1 | 12 | 13
  Stage III | 0 | 5 | 5
  Missing | 0 | 3 | 3
Eastern Cooperative Oncology Group performance status (ECOG P.S.) [Count of Participants; unit: Participants] — ECOG P.S.) assess participant's performance status on 5 point scale: 0=Fully active/able to carry on all pre-disease activities without restriction; 1=restricted in physically strenuous activity, ambulatory/able to carry out light or sedentary work; 2=ambulatory ( greater than [>] 50 percent [%] of waking hours), capable of all self-care, unable to carry out any work activities; 3=capable of only limited self-care, confined to bed/chair >50% of waking hours; 4=completely disabled, cannot carry on any self-care, totally confined to bed/chair; 5=dead.
  Participants
    Scale = 0 | 4 | 29 | 33
    Scale = 1 | 2 | 8 | 10
    Scale = 2 | 0 | 2 | 2
    Scale = 3 | 0 | 0 | 0
    Scale = 4 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS) Rate at 12 Months From the Start of Study Treatment
Description: PFS rate was defined as the percentage of participants who were alive and have not had disease progression at 12 months after the date of first dose of treatment in Treatment Period I. PFS was assessed by International Myeloma Working Group (IMWG) Criteria (2014 version). Per IMWG criteria, progressive disease (PD): serum M-component increase ≥0.5 g/dl or urine M-component increase ≥200 mg/24-hour/ difference between involved and uninvolved free light chain (FLC) levels increase >10 mg/dl or bone marrow plasma cell ≥10%/ development of new/ increase in size of existing bone lesions or soft tissue plasmacytoma or development of hypercalcemia.
Time Frame: Up to 12 months
Population: as for baseline characteristics
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Groups:
- [Overall]; Combination Therapy + Ixazomib Therapy: Bortezomib + Lenalidomide + Dexamethasone, or Carfilzomib + Lenalidomide + Dexamethasone, standard recommended dose according to the package insert of each drug (Treatment Period I), followed by Ixazomib (4.0 mg) on Days 1, 8 and 15, plus Lenalidomide (25 mg) on Days 1 to 21, and Dexamethasone (40 mg) on Days 1, 8, 15 and 22, of a 28-day cycle (Treatment Period II)
Arm/Group | [VRd]; Bortezomib + Lenalidomide + Dexamethasone Therapy | [KRd]; Carfilzomib + Lenalidomide + Dexamethasone Therapy | [Overall]; Combination Therapy + Ixazomib Therapy
Number analyzed (Participants) | 6 | 39 | 45
Percentage of Participants | 50.0 [15.3 to 84.7] | 48.7 [34.7 to 62.9] | 48.9 [35.9 to 62.0]

2. Secondary Outcome: Overall Survival (OS) From the Start of Study Treatment
Description: OS was defined as the period from the first dose of treatment in Treatment Period I to the time when death (regardless of the cause of death) was confirmed. Participants who were still alive were censored at the last confirmed date of survival or the date of data cut-off, whichever was earlier.
Time Frame: Up to 39 months as a maximum
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | [VRd]; Bortezomib + Lenalidomide + Dexamethasone Therapy | [KRd]; Carfilzomib + Lenalidomide + Dexamethasone Therapy | [Overall]; Combination Therapy + Ixazomib Therapy
Number analyzed (Participants) | 6 | 39 | 45
Months | NA [16.00 to NA] — NA: Data not available due to below the level of detection and insufficient number of participants with events. OS data were not mature, and the median OS was not reached. | NA [NA to NA] — NA: Data not available due to below the level of detection and insufficient number of participants with events. OS data were not mature, and the median OS was not reached. | NA [NA to NA] — NA: Data not available due to below the level of detection and insufficient number of participants with events. OS data were not mature, and the median OS was not reached.

3. Secondary Outcome: PFS From the Start of Study Treatment
Description: PFS was defined as the period from the first dose of treatment in Treatment Period I to the time of confirmed PD or confirmed death (regardless of the cause of death), whichever is earlier. PFS was assessed by IMWG Criteria.
Time Frame: Up to 39 months as a maximum
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | [VRd]; Bortezomib + Lenalidomide + Dexamethasone Therapy | [KRd]; Carfilzomib + Lenalidomide + Dexamethasone Therapy | [Overall]; Combination Therapy + Ixazomib Therapy
Number analyzed (Participants) | 6 | 39 | 45
Months | NA [4.86 to NA] — NA: data not available due to below the level of detection and insufficient number of participants with events. PFS data were not mature, and the median PFS was not reached. | 28.96 [21.32 to NA] — NA: data not available due to below the level of detection and insufficient number of participants with events. PFS data were not mature, and the median PFS was not reached. | 28.96 [21.32 to NA] — NA: data not available due to below the level of detection and insufficient number of participants with events. PFS data were not mature, and the median PFS was not reached.

4. Secondary Outcome: Percentage of Participants Who Achieved VGPR or Better (CR + VGPR)
Description: VGPR or better (CR + VGPR) were assessed by IMWG Criteria. Per IMWG criteria, PR (partial response): ≥50% reduction of serum M protein+reduction in 24-hour urinary M protein by ≥90%/ to <200 mg/24-hour or ≥50% decrease in difference between involved and uninvolved free light chain (FLC) levels/ ≥50% reduction in bone marrow plasma cells, if ≥30% at baseline/ ≥50% reduction in size of soft tissue plasmacytomas. VGPR (very good PR): serum+urine M-protein detectable by immunofixation but not on electrophoresis/ ≥90% reduction in serum M-protein+urine Mprotein level <100 mg/24-hour. CR (complete response): negative immunofixation on serum+urine+disappearance of soft tissue plasmacytomas+<5% plasma cells in bone marrow.
Time Frame: Up to 39 months as a maximum
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | [VRd]; Bortezomib + Lenalidomide + Dexamethasone Therapy | [KRd]; Carfilzomib + Lenalidomide + Dexamethasone Therapy | [Overall]; Combination Therapy + Ixazomib Therapy
Number analyzed (Participants) | 6 | 39 | 45
Percentage of Participants | 33.3 [4.3 to 77.7] | 43.6 [27.8 to 60.4] | 42.2 [27.7 to 57.8]

5. Secondary Outcome: Number of Participants With Minimal Residual Disease (MRD) Positive or Negative in Bone Marrow in Participants Who Achieved CR
Description: MRD was measured by the flow cytometry method using bone marrow aspiration. Reported data were numbers of participants with MRD positive and negative in bone marrow in participants who achieved CR. MRD positive was categorized into three sensitivity levels with the numbers of cells counted (10^-4 to - Max; 10^-5 to 10^-4; 10^-6 to 10^-5). MRD negativity is defined as absence of MRD and MRD positivity is defined as presence of MRD. If a participant is MRD-positive at their first evaluation and MRD-negative after re-examination, the participant will be considered to be MRD-negative. CR will be assessed by IMWG Criteria.
Time Frame: Up to 39 months as a maximum
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | [VRd]; Bortezomib + Lenalidomide + Dexamethasone Therapy | [KRd]; Carfilzomib + Lenalidomide + Dexamethasone Therapy | [Overall]; Combination Therapy + Ixazomib Therapy
Number analyzed (Participants) | 2 | 9 | 11
Participants
  Sensitivity Level; 10^-4=< - Max | 0 | 1 | 1
  Sensitivity Level; 10^-5=< - <10^-4 | 1 | 2 | 3
  Sensitivity Level; 10^-6=< - <10^-5 | 1 | 1 | 2
  Negative | 0 | 5 | 5

6. Secondary Outcome: Percentage of Participants Who Achieve or Maintain Any Best Response
Description: Best response is defined as the cumulative numbers of participants who achieve each level of best response including PR, VGPR and CR assessed with IMWG Criteria, after each cycle of treatment. Per IMWG criteria, PR (partial response): ≥50% reduction of serum M protein+reduction in 24-hour urinary M protein by ≥90%/ to <200 mg/24-hour or ≥50% decrease in difference between involved and uninvolved free light chain (FLC) levels/ ≥50% reduction in bone marrow plasma cells, if ≥30% at baseline/ ≥50% reduction in size of soft tissue plasmacytomas. VGPR (very good PR): serum+urine M-protein detectable by immunofixation but not on electrophoresis/ ≥90% reduction in serum M-protein+urine Mprotein level <100 mg/24-hour. CR (complete response): negative immunofixation on serum+urine+disappearance of soft tissue plasmacytomas+<5% plasma cells in bone marrow.
Time Frame: Up to 39 months as a maximum
Population: as for baseline characteristics
Measure: Number; unit: Percentage of Participants
Arm/Group | [VRd]; Bortezomib + Lenalidomide + Dexamethasone Therapy | [KRd]; Carfilzomib + Lenalidomide + Dexamethasone Therapy | [Overall]; Combination Therapy + Ixazomib Therapy
Number analyzed (Participants) | 6 | 39 | 45
Percentage of Participants
  CR | 33.3 | 23.1 | 24.4
  VGPR | 0 | 20.5 | 17.8
  PR | 50.0 | 28.2 | 31.1

7. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR is defined as the percentage of participants who achieve a best response of PR or better including stringent complete response (sCR), VGPR and PR assessed with IMWG Criteria, after the start of the study treatment. Per IMWG criteria, PR (partial response): ≥50% reduction of serum M protein+reduction in 24-hour urinary M protein by ≥90%/ to <200 mg/24-hour or ≥50% decrease in difference between involved and uninvolved free light chain (FLC) levels/ ≥50% reduction in bone marrow plasma cells, if ≥30% at baseline/ ≥50% reduction in size of soft tissue plasmacytomas. VGPR (very good PR): serum+urine M-protein detectable by immunofixation but not on electrophoresis/ ≥90% reduction in serum M-protein+urine Mprotein level <100 mg/24-hour. CR (complete response): negative immunofixation on serum+urine+disappearance of soft tissue plasmacytomas+<5% plasma cells in bone marrow.
Time Frame: Up to 39 months as a maximum
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | [VRd]; Bortezomib + Lenalidomide + Dexamethasone Therapy | [KRd]; Carfilzomib + Lenalidomide + Dexamethasone Therapy | [Overall]; Combination Therapy + Ixazomib Therapy
Number analyzed (Participants) | 6 | 39 | 45
Percentage of Participants | 83.3 [35.9 to 99.6] | 71.8 [55.1 to 85.0] | 73.3 [58.1 to 85.4]

8. Secondary Outcome: Percentage of Participants Continuing Treatment With Ixazomib at 12 Months From the Start of Study Treatment
Time Frame: 12 months
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | [VRd]; Bortezomib + Lenalidomide + Dexamethasone Therapy | [KRd]; Carfilzomib + Lenalidomide + Dexamethasone Therapy | [Overall]; Combination Therapy + Ixazomib Therapy
Number analyzed (Participants) | 6 | 39 | 45
Percentage of Participants | 50.0 [11.8 to 88.2] | 35.9 [21.2 to 52.8] | 37.8 [23.8 to 53.5]

9. Secondary Outcome: Duration of Response (DOR)
Description: DOR is defined as the time from the date of first documentation of response ≥PR to the date of first documentation of PD or death due to any cause. PR and PD will be assessed with IMWG Criteria. Per IMWG criteria, PR (partial response): ≥50% reduction of serum M protein+reduction in 24-hour urinary M protein by ≥90%/ to <200 mg/24-hour or ≥50% decrease in difference between involved and uninvolved free light chain (FLC) levels/ ≥50% reduction in bone marrow plasma cells, if ≥30% at baseline/ ≥50% reduction in size of soft tissue plasmacytomas. VGPR (very good PR): serum+urine M-protein detectable by immunofixation but not on electrophoresis/ ≥90% reduction in serum M-protein+urine Mprotein level <100 mg/24-hour. CR (complete response): negative immunofixation on serum+urine+disappearance of soft tissue plasmacytomas+<5% plasma cells in bone marrow.
Time Frame: Up to 39 months as a maximum
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | [VRd]; Bortezomib + Lenalidomide + Dexamethasone Therapy | [KRd]; Carfilzomib + Lenalidomide + Dexamethasone Therapy | [Overall]; Combination Therapy + Ixazomib Therapy
Number analyzed (Participants) | 5 | 28 | 33
Months | 15.31 [3.64 to NA] — NA: data not available due to below the level of detection and insufficient number of participants with events. DOR data were not mature. | 28.03 [20.4 to NA] — NA: data not available due to below the level of detection and insufficient number of participants with events. DOR data were not mature. | 28.03 [20.4 to NA] — NA: data not available due to below the level of detection and insufficient number of participants with events. DOR data were not mature.

10. Secondary Outcome: Time to Next Treatment (TTNT)
Description: TTNT is defined as the period from the start of study treatment Period I to the start of next line treatment.
Time Frame: Up to 39 months as a maximum
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | [VRd]; Bortezomib + Lenalidomide + Dexamethasone Therapy | [KRd]; Carfilzomib + Lenalidomide + Dexamethasone Therapy | [Overall]; Combination Therapy + Ixazomib Therapy
Number analyzed (Participants) | 6 | 39 | 45
Months | 21.59 [4.99 to NA] — NA: Upper limit for 95% CI was not available due to below the level of detection and insufficient number of participants with events. | 32.26 [12.43 to 35.44] | 32.26 [14.88 to 35.44]

11. Secondary Outcome: Duration of Therapy (DOT)
Description: DOT is defined as the treatment duration of study drug at study treatment Period I.
Time Frame: Up to 39 months as a maximum
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | [VRd]; Bortezomib + Lenalidomide + Dexamethasone Therapy | [KRd]; Carfilzomib + Lenalidomide + Dexamethasone Therapy | [Overall]; Combination Therapy + Ixazomib Therapy
Number analyzed (Participants) | 6 | 39 | 45
Months | 14.69 [4.86 to NA] — NA: Upper limit for 95% CI was not available due to below the level of detection and insufficient number of participants with events. | 12.43 [7.74 to 24.79] | 12.43 [8.86 to 24.79]

12. Secondary Outcome: Patient-Reported Outcome Health-Related Quality of Life (HRQoL) Based on Global Health Status Scale of European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-C30 (EORTC QLQ-C30)
Description: EORTC QLQ-C30 contains 30 items across 5 functional scales (physical, role, cognitive, emotional, and social), 9 symptom scales (fatigue, nausea and vomiting, pain, dyspnea, sleep disturbance, appetite loss, constipation, diarrhea, and financial difficulties) and a global health status/QOL scale (Global Health Status). EORTC QLQ-C30 contains 28 questions (4-point scale where 1=Not at all [best] to 4=Very Much [worst]) and 2 questions (7-point scale where 1=Very poor [worst] to 7= Excellent [best]). Raw scores are converted into scale scores ranging from 0 to 100. For the functional scales and the global health status/QOL scale, higher scores represent better QOL; for the symptom scales, lower scores represent better QOL.
Time Frame: Baseline and End of Treatment (Up to 23 cycles for VRd Group, Up to 32 cycles for KRd and Overall Group, each cycle was of 28 days)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | [VRd]; Bortezomib + Lenalidomide + Dexamethasone Therapy | [KRd]; Carfilzomib + Lenalidomide + Dexamethasone Therapy | [Overall]; Combination Therapy + Ixazomib Therapy
Number analyzed (Participants) | 6 | 39 | 45
Score on a Scale
  Baseline | 44.44 (40.369) | 63.25 (24.085) | 60.74 (26.981)
  Cycle 23: number analyzed (Participants) | 1 | 6 | 7
  Cycle 23 | 0 (NA) — NA: data not available due to below the level of detection and insufficient number of participants with events. | 54.17 (8.740) | 46.43 (21.973)
  Cycle 32: number analyzed (Participants) | 0 | 2 | 2
  Cycle 32 |  | 50.00 (23.750) | 50.00 (23.750)

13. Secondary Outcome: Patient-Reported Outcome HRQoL Based on EORTC Multiple Myeloma Module (EORTC QLQ-MY20) Score
Description: EORTC QLQ-MY20 has 20 items across 4 independent subscales, 2 functional subscales (body image, future perspective), and 2 symptoms scales (disease symptoms, and side effects of treatment). Scores are averaged, and transformed to 0-100 scale. For the functional scales, high scores represent improvement. For the symptom scales, higher scores represent worsening.
Time Frame: as for outcome 12
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | [VRd]; Bortezomib + Lenalidomide + Dexamethasone Therapy | [KRd]; Carfilzomib + Lenalidomide + Dexamethasone Therapy | [Overall]; Combination Therapy + Ixazomib Therapy
Number analyzed (Participants) | 6 | 39 | 45
Score on a Scale
  Disease Symptoms: Baseline | 24.07 (21.564) | 19.23 (16.756) | 19.88 (17.266)
  Disease Symptoms: Cycle 23: number analyzed (Participants) | 1 | 6 | 7
  Disease Symptoms: Cycle 23 | 0 (NA) — Number of participants analyzed was one. | 4.63 (7.384) | 3.97 (6.964)
  Disease Symptoms: Cycle 32: number analyzed (Participants) | 0 | 2 | 2
  Disease Symptoms: Cycle 32 |  | 2.78 (3.928) | 2.78 (3.928)
  Side-Effects of Treatment: Baseline | 16.67 (12.776) | 16.60 (14.464) | 16.61 (14.115)
  Side-Effects of Treatment: Cycle 23: number analyzed (Participants) | 1 | 6 | 7
  Side-Effects of Treatment: Cycle 23 | 3.70 (NA) — Number of participants analyzed was one. | 16.05 (3.825) | 14.29 (5.828)
  Side-Effects of Treatment: Cycle 32: number analyzed (Participants) | 0 | 2 | 2
  Side-Effects of Treatment: Cycle 32 |  | 18.52 (15.713) | 18.52 (15.713)
  Body Image: Baseline | 44.44 (45.542) | 23.08 (26.660) | 25.93 (30.058)
  Body Image: Cycle 23: number analyzed (Participants) | 1 | 6 | 7
  Body Image: Cycle 23 | 0 (NA) — Number of participants analyzed was one. | 16.67 (18.257) | 14.29 (17.817)
  Body Image: Cycle 32: number analyzed (Participants) | 0 | 2 | 2
  Body Image: Cycle 32 |  | 16.67 (23.570) | 16.67 (23.570)
  Future Perspective: Baseline | 66.67 (37.185) | 44.16 (24.114) | 47.16 (26.817)
  Future Perspective: Cycle 23: number analyzed (Participants) | 1 | 6 | 7
  Future Perspective: Cycle 23 | 11.11 (NA) — Number of participants analyzed was one. | 35.19 (8.364) | 31.75 (11.878)
  Future Perspective: Cycle 32: number analyzed (Participants) | 0 | 2 | 2
  Future Perspective: Cycle 32 |  | 27.78 (7.857) | 27.78 (7.857)

14. Secondary Outcome: Evaluation of Modified Quality-Adjusted Life-Years (QALYs)
Description: Modified QALYs was calculated from the score of EORTC QLQ-C30. The health-related quality of life scale score of EORTC QLQ-C30 was converted into a utility value ranging from 0 (dead) to 1 (perfect health), and used to adjust the value of survival years; this value was assessed as the modified QALY.
Time Frame: Up to 39 months as a maximum
Population: as for baseline characteristics
Measure: Median (Full Range); unit: Quality-Adjusted Life-Years
Arm/Group | [VRd]; Bortezomib + Lenalidomide + Dexamethasone Therapy | [KRd]; Carfilzomib + Lenalidomide + Dexamethasone Therapy | [Overall]; Combination Therapy + Ixazomib Therapy
Number analyzed (Participants) | 4 | 16 | 20
Quality-Adjusted Life-Years | 0.467 [0.25 to 0.89] | 0.534 [0.17 to 0.85] | 0.518 [0.17 to 0.89]

15. Secondary Outcome: Healthcare Resource Utilization (HCRU): Number of Events With Hospitalization Per Participants-Month
Description: HCRU was calculated from Exposure-adjusted rate of hospitalization events (per participants-months) and the duration of hospitalization among participants in Treatment Period I and Treatment Period II. Number of events with hospitalization per participants-month in Treatment Period I and Treatment Period II was reported.
Time Frame: Up to 39 months as a maximum
Population: as for baseline characteristics
Measure: Number; unit: Number of Events per Participants-Month
Arm/Group | [VRd]; Bortezomib + Lenalidomide + Dexamethasone Therapy | [KRd]; Carfilzomib + Lenalidomide + Dexamethasone Therapy | [Overall]; Combination Therapy + Ixazomib Therapy
Number analyzed (Participants) | 6 | 39 | 45
Number of Events per Participants-Month | 1.9 | 2.9 | 2.7

16. Secondary Outcome: Healthcare Resource Utilization (HCRU): Duration of Hospital Stay Per Participants
Description: HCRU was calculated from Exposure-adjusted rate of hospitalization events (per participants-months) and the duration of hospitalization among participants in Treatment Period I and Treatment Period II. Duration of hospital stay per participants in Treatment Period I and Treatment Period II was reported.
Time Frame: Up to 39 months as a maximum
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | [VRd]; Bortezomib + Lenalidomide + Dexamethasone Therapy | [KRd]; Carfilzomib + Lenalidomide + Dexamethasone Therapy | [Overall]; Combination Therapy + Ixazomib Therapy
Number analyzed (Participants) | 6 | 39 | 45
Days | 14.8 (16.01) | 19.4 (18.14) | 18.8 (17.77)

17. Secondary Outcome: Relative Dose Intensity (RDI)
Description: RDI for each study drug is defined as 100*(Total amount of dose taken)/(Total prescribed dose of treated cycles), where total prescribed dose equals [dose prescribed at enrollment* number of prescribed doses per cycle* the number of treated cycles].
Time Frame: Up to 39 months as a maximum
Population: as for baseline characteristics
Measure: Median (Full Range); unit: Percent
Arm/Group | [Overall]; Combination Therapy + Ixazomib Therapy
Number analyzed (Participants) | 45
Percent
  Bortezomib, Ixazomib: number analyzed (Participants) | 6
  Bortezomib, Ixazomib | 71.93 [58.2 to 97.2]
  Carfilzomib, Ixazomib: number analyzed (Participants) | 39
  Carfilzomib, Ixazomib | 87.70 [27.0 to 108.4]
  Bortezomib/Carfilzomib, Ixazomib | 83.24 [27.0 to 108.4]
  Lenalidomide | 47.18 [9.0 to 100.4]
  Dexamethasone | 48.61 [6.6 to 105.3]

18. Secondary Outcome: Percentage of Participants With Bone Lesions (Bone Evaluation)
Time Frame: Up to 39 months as a maximum
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | [VRd]; Bortezomib + Lenalidomide + Dexamethasone Therapy | [KRd]; Carfilzomib + Lenalidomide + Dexamethasone Therapy | [Overall]; Combination Therapy + Ixazomib Therapy
Number analyzed (Participants) | 6 | 39 | 45
Percentage of Participants | 100.0 [29.2 to 100.0] | 59.1 [36.4 to 79.3] | 64.0 [42.5 to 82.0]

19. Secondary Outcome: Number of Participants Reporting One or More Treatment-Emergent AEs (TEAEs)
Description: An adverse event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. A TEAE is defined as an adverse event with an onset that occurs after receiving study drug.
Time Frame: Up to 39 months as a maximum
Population: Safety Analysis Set: all participants who were enrolled in Treatment Period I and who receive at least one dose of any therapy during the Treatment Period.
Measure: Count of Participants; unit: Participants
Arm/Group | [VRd]; Bortezomib + Lenalidomide + Dexamethasone Therapy | [KRd]; Carfilzomib + Lenalidomide + Dexamethasone Therapy | [Overall]; Combination Therapy + Ixazomib Therapy
Number analyzed (Participants) | 6 | 39 | 45
Participants | 6 | 35 | 41

ADVERSE EVENTS:
Time Frame: Up to 39 months as a maximum
Description: At each visit the investigator had to document any occurrence of adverse events (AEs) and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment. In this study, only AEs in total duration of both Treatment Period I and II were planned to be collected on the study protocol and reported in this section. There were no plans to collect AEs for each Period.
Arm/Group | [VRd]; Bortezomib + Lenalidomide + Dexamethasone Therapy | [KRd]; Carfilzomib + Lenalidomide + Dexamethasone Therapy | [Overall]; Combination Therapy + Ixazomib Therapy
All-Cause Mortality (participants affected / at risk) | 0/6 | 2/39 | 2/45
Serious Adverse Events (participants affected / at risk) | 3/6 | 14/39 | 17/45
Other Adverse Events (participants affected / at risk) | 6/6 | 31/39 | 37/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | [VRd]; Bortezomib + Lenalidomide + Dexamethasone Therapy (N=6) | [KRd]; Carfilzomib + Lenalidomide + Dexamethasone Therapy (N=39) | [Overall]; Combination Therapy + Ixazomib Therapy (N=45)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 1
Prinzmetal angina (Cardiac disorders) | 0 | 1 | 1
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1 | 1
Enterocolitis (Gastrointestinal disorders) | 0 | 1 | 1
Pyrexia (General disorders) | 0 | 1 | 1
Bile duct stone (Hepatobiliary disorders) | 0 | 1 | 1
Pneumonia (Infections and infestations) | 0 | 5 | 5
Influenza (Infections and infestations) | 0 | 2 | 2
Gastroenteritis (Infections and infestations) | 0 | 1 | 1
Pneumonia bacterial (Infections and infestations) | 0 | 1 | 1
Compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 1 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 2 | 2
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | [VRd]; Bortezomib + Lenalidomide + Dexamethasone Therapy (N=6) | [KRd]; Carfilzomib + Lenalidomide + Dexamethasone Therapy (N=39) | [Overall]; Combination Therapy + Ixazomib Therapy (N=45)
Anaemia (Blood and lymphatic system disorders) | 1 | 3 | 4
Diarrhoea (Gastrointestinal disorders) | 3 | 10 | 13
Constipation (Gastrointestinal disorders) | 1 | 3 | 4
Malaise (General disorders) | 1 | 3 | 4
Pyrexia (General disorders) | 1 | 3 | 4
Nasopharyngitis (Infections and infestations) | 2 | 2 | 4
White blood cell count decreased (Investigations) | 2 | 9 | 11
Platelet count decreased (Investigations) | 1 | 8 | 9
Neutrophil count decreased (Investigations) | 1 | 6 | 7
Decreased appetite (Metabolism and nutrition disorders) | 3 | 0 | 3
Taste disorder (Nervous system disorders) | 2 | 1 | 3
Rash (Skin and subcutaneous tissue disorders) | 4 | 3 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2019-05-30): https://cdn.clinicaltrials.gov/large-docs/74/NCT03416374/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-01): https://cdn.clinicaltrials.gov/large-docs/74/NCT03416374/SAP_001.pdf